CLINICAL TRIAL: NCT03518463
Title: Enhanced Recovery After Surgery Versus Standard Recovery for Emergency Caesarean Deliveries at Mbarara Hospital, Uganda: A Randomized Control Trial
Brief Title: Enhanced Recovery After Surgery for Emergency Caesarean Deliveries
Acronym: ERAS-Mbarara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUST 0606/2018
Record Dates: First submitted 2018-04-16; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: The ERAS arm was exposed to modified ERAS elements including preoperative counseling and education, prophylaxis against nausea and vomiting (PONV), individualized goal directed fluid therapy, early mobilization at 6-8 hours postoperative, early feeding within 1 hour postoperative,urethral catheter removal at 6 hours, oral fixed combination non opioid analgesia, oral antibiotics and anti-emetics. PONV included intravenous metoclopromide and dexametasone, no ondansetron given. Patients in the control arm recovered with routine care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Mothers delivering by emergency CS were randomly assigned to either ERAS or routine care arms in a ratio of 1:1. We did simple randomization to either ERAS or routine care arm without any blocks. We generated patient group assignments using the computer algorithm (computer-generated list of random numbers) and placed in identical sealed opaque envelopes. A statistician not involved in the research generated the random number list. The envelopes were opened sequentially by the anesthetist when an eligible patient was encountered. Mothers were recruited into the study by the two research assistants implementing ERAS elements. Single blinding of PI and the two research assistants assessing outcomes was done to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): ERAS arm received;
  Preoperative:1. Intravenous (IV) cefazoline 1g 2. IV metoclopromide 10mg, dexamethasone 8mg, ranitidine 150mg
  Intraoperative: 1. Hyperbaric bupivacaine 10-15mg plus intrathecal morphine 100mcg 2. Adrenaline 100mcg in 500ml of ringers lactate 3. Individualized goal directed fluid therapy 4. Reinforced counseling and education 5. wound infiltration with isobaric bupivacaine 2mg/kg 6. Rectal diclofenac 100mg and misoprostol 400mcg stat
  Postoperative:
  1. Feeding within 1 hour
  2. urethral catheter removal at 6-8 hours
  3. Mobilization at 8-10 hours
  4. A single fixed dose combination of ibuprofen 400 mg and paracetamol 500 mg 8 hourly
  5. Tablets Amoxicillin-clavulunate 850mg 12 hourly
  Interventions: Combination Product: Enhanced recovery after surgery (ERAS)
- Control (Active Comparator): Standard care arm received;
  1. IV ceftriaxone 2g or ampiclox 2g
  2. Anesthetists administered IV fluids, vasopressors, and managed hypothermia based on their clinical impressions.
  3. Oral feeding and breastfeeding were allowed any time after transfer to postnatal ward.
  4. Urethral catheters were removed between 12-24 hours after surgery.
  5. Ward nurses and obstetricians made decisions regarding treatment without study staff input or oversight.
  Interventions: Combination Product: Enhanced recovery after surgery (ERAS)

INTERVENTIONS:
Combination Product: Enhanced recovery after surgery (ERAS) — The ERAS arm was exposed to standard preoperative, intraoperative and postoperative ERAS protocols of care. However, some were modified to our local resources and requirements as well as to the emergency nature of the surgeries.
  Other Names: Accelerated recovery; Fast track surgery

SUMMARY:
Caesarean section (CS) constitutes a large proportion of the total surgical volume in low-income countries. This rate comes with challenges including surgical complications, shortage of beds, and consequently long waiting time for operations and high costs. These have led to the adoption of ERAS in developed countries in a bid to save costs by reducing hospital length of stay without compromising the health of the mother and her baby.

DETAILED DESCRIPTION:
CS is the most common major surgery at Mbarara Hospital (56.2%). This rate comes with challenges including surgical complications, shortage of beds, and consequently long waiting time for operations. Enhanced recovery programs are composed of preoperative, intraoperative and postoperative strategies combined to form a multi-modal pathway. ERAS requires a multidisciplinary team of anesthetists, surgeons and nurses for successful implementation and realization of its advantages. ERAS has been seen to reduce duration of hospital stay, complications and costs. Although many of the elements of enhanced recovery after surgery are similar, it has not been tested in emergency CS and there is limited data about its applicability in low income settings like Uganda where 95% of CS are emergencies. The aim of this study was to assess the impact of ERAS protocols following emergency caesarean delivery in a low resource setting.

ELIGIBILITY:
Inclusion Criteria:

* We included women who were ASA 1 and 2 mothers who were delivering by emergency caesarean section using spinal anesthetic technique.

Exclusion Criteria:

* Exclusion criteria included refusal to consent, pregnancy complicated by preeclampsia, antepartum hemorrhage, malaria, gestational diabetes mellitus, physical disability that would prevent postoperative mobilization and mental illness precluding comprehension of protocols.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All pregnant mothers with whom a decision to deliver by emergency caesarean section has been made
Enrollment: 160 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Measured from surgery up to 120 hours.
  Length of hospital stay was measured in hours

SECONDARY OUTCOMES:
Complication rates | Pain was assessed after 6 hours postoperative; PONV, pruritus and urine retention were assessed for 24 hours; headache was assessed for 1 week; wound infection, puerperal sepsis and readmission were assessed up to 30 days postoperative
  These included pain, PONV, headache, pruritus, urine retention, wound infection, puerperal sepsis and readmission

CONTACTS AND LOCATIONS:
Overall Officials: Baluku Moris, MD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara university of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after obtaining all necessary permission.